CLINICAL TRIAL: NCT07193563
Title: The ENCalmSocial Trial: A Randomized, Double-Blind, Placebo-Controlled Monotherapy Trial to Evaluate the Efficacy and Safety of ENX-102 in Participants With Social Anxiety Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of ENX-102 in Participants With Social Anxiety Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Engrail Therapeutics INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENX-102-005
Record Dates: First submitted 2025-09-24; First posted 2025-09-26 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Social Anxiety Disorder (SAD)
Keywords: Social Anxiety; ENX-102
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ENX-102 (Experimental): Participants will receive 2 mg of ENX-102 in capsule form orally once daily for 6 weeks, followed by 2 weeks of tapered dose and up to 2 weeks of placebo in capsule form before and/or after the 8-week ENX-102 treatment period.
  Interventions: Drug: ENX-102
- Placebo (Placebo Comparator): Participants will receive ENX-102 matching placebo in capsule once daily for 10 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ENX-102 — oral capsule
  Arms: ENX-102
Other: Placebo — oral capsule
  Arms: Placebo

SUMMARY:
This is a double-blind study to evaluate the efficacy and safety of ENX-102 in participants with social anxiety disorder (SAD).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female at birth, aged 18-70 years, inclusive, at screening Diagnosed with SAD according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR), confirmed by a Mini-International Neuropsychiatric Interview (MINI) version 7.0.2
* LSAS total score of ≥70
* CGI-S score of ≥4

Key Exclusion Criteria:

* Clinically predominant psychiatric diagnosis other than SAD per the MINI
* Any past/lifetime or current diagnosis of a neurocognitive disorder or psychotic disorder, or any current diagnosis of posttraumatic stress disorder, obsessive compulsive disorder, or bipolar disorder
* Reports moderately severe to severe symptoms of depression
* Frequent use of benzodiazepines within 90 days of screening
* Used prohibited medication or prohibited herbal or other supplements within 5 half- lives or 21 days prior to Day 1 and unwillingness to refrain from their use for the duration of the trial
* Recent suicidal ideation or behavior
* Current or recent moderate or severe substance use disorder as assessed by the MINI
* Is unwilling/unable to abstain from alcohol, marijuana, THC, CBD, and/or any other psychoactive substances (except for nicotine or caffeine) for the duration of the trial, per Investigator judgment, and/or has a positive alcohol test or drug test at Screening or Day 1
* Clinically significant abnormal findings in safety assessments
* Has significant progressive disorders or unstable medical conditions Unable to comply with the requirements of the study or, in the opinion of the Investigator or Sponsor, is unsuitable for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline on the Clinician-administered Liebowitz Social Anxiety Scale (LSAS) - Total score | Baseline (Day 1) and Week 6
  The LSAS is a 24-item semi-structured interview measure of fear and avoidance experienced in a range of social and performance situations. The 24 items are divided into 2 subscales, 13 concerning performance anxiety & 11 pertaining to social situations. The 24 items are first rated on a Likert Scale from 0 to 3 on fear felt during the situations (0=none, 1=mild, 2=moderate, 3= severe), and then the same items are rated regarding avoidance of the situation (0=never, 1=occasionally, 2=often, 3=usually). An overall global score (0 to 144) is calculated by adding total fear/anxiety and total avoidance scores. Higher scores indicated higher probability of social anxiety disorder.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - IMA Clinical Research Phoenix, Phoenix, Arizona
  - University of California, La Jolla, California
  - Neuroresearch Group, Los Angeles, California
  - Excell Research, Inc., Oceanside, California
  - Anderson Clinical Research, Redlands, California
  - California Neuroscience Research, LLC, Sherman Oaks, California
  - Sunwise Clincial Research, Walnut Creek, California
  - Mountain View Clinical Research, Denver, Colorado
  - CNS Health, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - CenExel iResearch, LLC, Savannah, Georgia
  - IMA Clinical Research, Las Vegas, Nevada
  - Redbird Research, Las Vegas, Nevada
  - Cenexel HRI, Berlin, New Jersey
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Clinical Neurosciences, Inc, Memphis, Tennessee
  - Austin Clinical Trials Partners, Austin, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: No